CLINICAL TRIAL: NCT02463097
Title: Safety Evaluation of the Hybrid Closed Loop (HCL) System in Type 1 Diabetes
Brief Title: Hybrid Closed Loop Pivotal Trial in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 294
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): All subjects wearing the MMT-670G insulin pump, using it with the closed loop algorithm
  Interventions: Device: Insulin Pump

INTERVENTIONS:
Device: Insulin Pump — Closed Loop Algorithm
  Other Names: MMT-670G

SUMMARY:
This study is a single-arm, multi-center, Home and Hotel Clinical Investigation in subjects with type 1 diabetes on insulin pump therapy. The purpose of this study is to demonstrate that the closed loop algorithm that is built into the 670G insulin pump is safe as part of the overall system.

DETAILED DESCRIPTION:
The study will proceed as follows:

Run-in Period:

A total of up to 150 subjects (age 14 - 75) will be enrolled at up to 10 investigational centers (9 in the US, 1 in the Europe, Middle East and Africa (EMEA) region) in order to reach 100 subjects who will complete the HCL study. The 2-week run-in period will be used to allow subjects to become familiar with new study devices. During the two week run-in period subjects will be using the Study Pump (670G) with the Sensor Augmented Pump function only activated (i.e. SmartGuard OFF and HCL OFF).

Study Period - At Home:

Following the two week run-in period using the Study Pump (670G), all subjects will participate in a 3-month study period.

Subjects will be required to have a companion with them during the night for the duration of the study period. Companions will need to be under the same roof, but not necessarily in the same bedroom. During the Hotel stay where subjects are monitored closely, the presence of a companion is not necessary.

Study Period - Hotel Study Subjects will participate in a Hotel study (6 days, 5 nights), with the remainder of the study period to be spent at home.

All subjects will undergo daytime and nighttime Frequent Sample Testing (FST) for approximately 24 hours during the Hotel study with YSI or i-STAT® used as a reference value.

With respect to meals, subjects will be allowed to eat as they normally do.

Continued Access Program Subjects will be given the opportunity to extend use of their study devices for a period of 3 years. If subjects choose to participate in the continuation period, they will retain the study devices at the end of study period visit or receive them back in the event they have been returned to study staff already. During the continuation period, subjects will come in for office visits every 3 months. At each of the quarterly visits, subjects will be asked about the occurrence of adverse events and device complaints.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 14 - 75 years at time of screening
2. Has a clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Is willing to participate in a hotel study for the specified duration of hotel stay.
4. Must have companion who will sleep in the same dwelling place every night during the study period and should also be able to call the subject daily in the event the subject is traveling.
5. Is willing to perform ≥ 4 finger stick blood glucose measurements daily
6. Is willing to perform required sensor calibrations
7. Is willing to wear the system continuously throughout the study
8. Has a Glycosylated hemoglobin (A1C) value less than 10.0% (as processed by Central Lab) at time of screening visit
9. Has TSH in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
10. Pump therapy for greater than 6 months prior to screening (with or without CGM experience)
11. Is willing to upload data from the study pump, must have Internet access and a computer system that meets the requirements for uploading the study pump
12. If subject has celiac disease, it has been adequately treated as determined by the investigator
13. Is willing to take one of the following insulins and can financially support the use of either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount)

    * Humalog® (insulin lispro injection)
    * NovoLog® (insulin aspart)
14. With history of cardiovascular event 1 year or more from the time of screening must have an EKG within 6 months prior to screening or during screening. If subject has an abnormal EKG, participation is allowed if there is clearance from a cardiologist
15. With 3 or more cardiovascular risk factors listed below must have an EKG within 6 months prior to screening or during screening. If subject has an abnormal EKG, participation is allowed if there is clearance from a cardiologist

    Cardiovascular risk factors include:
    * Age >35 years
    * Type 1 diabetes of >15 years' duration
    * Presence of any additional risk factor for coronary artery disease
    * Presence of microvascular disease (proliferative retinopathy or nephropathy, including microalbuminuria)
    * Presence of peripheral vascular disease
    * Presence of autonomic neuropathy
16. With history of cardiovascular event 1 year or more from the time of screening must have a stress test within 6 months prior to screening or during run in period. If subject fails stress test, participation is allowed if there is clearance from a cardiologist
17. Must be able to speak and be literate in English

Exclusion Criteria:

1. Has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:

   * Medical assistance (i.e. Paramedics, Emergency Room ( ER) or Hospitalization)
   * Coma
   * Seizures
2. Is unable to tolerate tape adhesive in the area of sensor placement
3. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
4. Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
5. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
6. Is being treated for hyperthyroidism at time of screening
7. Has diagnosis of adrenal insufficiency
8. Has had DKA in the 6 months prior to screening visit.
9. Has taken any oral, injectable, or intravenous (IV) steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study
10. Actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
11. Has been hospitalized or has visited the ER in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes
12. Currently abusing illicit drugs
13. Currently abusing marijuana.
14. Currently abusing prescription drugs
15. Currently abusing alcohol
16. Using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening
17. Has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
18. Has elective surgery planned that requires general anesthesia during the course of the study
19. Has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
20. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation
21. Diagnosed with current eating disorder such as anorexia or bulimia
22. Diagnosed with chronic kidney disease that results in chronic anemia
23. Hematocrit that is below the normal reference range of lab used.
24. On dialysis
25. Serum creatinine of >2 mg/dL.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - AMCR Institute, Escondido, California
  - Stanford University Medical Center, Palo Alto, California
  - Barbara Davis Center for Childhood Diabetes (Adult), Aurora, Colorado
  - Barbara Davis Center for Childhood Diabetes (Pediatric), Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Park Nicollet Clinic-International Diabetes Center - Adult and Pediatric, Minneapolis, Minnesota
  - University of Virginia, Charlottesville, Virginia
  - Rainer Clinical Research Center, Renton, Washington
- Institute of Endocrinology, Sheba Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Cordero TL, Garg SK, Brazg R, Bailey TS, Shin J, Lee SW, Kaufman FR. The Effect of Prior Continuous Glucose Monitoring Use on Glycemic Outcomes in the Pivotal Trial of the MiniMed 670G Hybrid Closed-Loop System. Diabetes Technol Ther. 2017 Dec;19(12):749-752. doi: 10.1089/dia.2017.0208. Epub 2017 Nov 17. PMID 29148821
- [Derived] Garg SK, Weinzimer SA, Tamborlane WV, Buckingham BA, Bode BW, Bailey TS, Brazg RL, Ilany J, Slover RH, Anderson SM, Bergenstal RM, Grosman B, Roy A, Cordero TL, Shin J, Lee SW, Kaufman FR. Glucose Outcomes with the In-Home Use of a Hybrid Closed-Loop Insulin Delivery System in Adolescents and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2017 Mar;19(3):155-163. doi: 10.1089/dia.2016.0421. Epub 2017 Jan 30. PMID 28134564

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: All subjects wearing the MMT-670G insulin pump, using it with the closed loop algorithm
  Insulin Pump: Closed Loop Algorithm
  i-STAT blood testing: Intravenous i-STAT blood testing is used for reference validation
  Blood Glucose Meter testing: Frequent finger stick blood glucose testing using a Blood Glucose meter is required
Period: Overall Study
Arm/Group | Study Arm
Started | 124
Completed | 123
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects wearing the MMT-670G insulin pump, using it with the closed loop algorithm.
Arm/Group | Study Arm
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 96
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (16.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 55
Region of Enrollment [Number; unit: participants]
  United States | 112
  Israel | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in A1C
Description: There is no statistically powered primary endpoint in this study. However, there will be a descriptive analysis of change in A1C.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Study Arm
Number analyzed (Participants) | 123
Percent | -0.5 (0.6)

2. Secondary Outcome: Number of Severe Hypoglycemia Events
Description: There is no statistically powered secondary endpoint in this study. However, there will be a descriptive analysis of the number of Severe Hypoglycemia events.
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | Study Arm
Number analyzed (Participants) | 124
events | 0

3. Secondary Outcome: Number of Diabetic Ketoacidosis (DKA) Events
Description: There is no statistically powered secondary endpoint in this study. However, there will be a descriptive analysis on number of Diabetic Ketoacidosis (DKA) Event.
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | Study Arm
Number analyzed (Participants) | 124
events | 0

ADVERSE EVENTS:
Time Frame: 3 Month
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/124
Serious Adverse Events (participants affected / at risk) | 2/124
Other Adverse Events (participants affected / at risk) | 66/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=124)
Appendicitis (Infections and infestations) | 1 (1)
Bacterial arthritis of right wrist (Infections and infestations) | 1 (1)
C-difficile diarrhea (Investigations) | 1 (1)
Worsening Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=124)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain for few days (Gastrointestinal disorders) | 1 (1)
Abrasion to left great toe (Injury, poisoning and procedural complications) | 1 (1)
Acute frontal sinusitis (Infections and infestations) | 1 (1)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacterial conjunctivitis (Infections and infestations) | 1 (1)
Benign paroxysmal positional vertigo (Ear and labyrinth disorders) | 1 (1)
Bicycle injury (Injury, poisoning and procedural complications) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cold (Infections and infestations) | 4 (5)
Cold-upper respiratory (Infections and infestations) | 1 (1)
Common cold (Infections and infestations) | 5 (5)
Conjunctivitis (Eye disorders) | 1 (1)
Cracked ulna (Injury, poisoning and procedural complications) | 1 (1)
Deviated septum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1)
Gastro pain (upset stomach), nausea (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Gastrointestinal virus (Infections and infestations) | 1 (1)
Head cold (Infections and infestations) | 3 (3)
Headache (Nervous system disorders) | 4 (5)
Heart burn (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
Infiltration. bruising. (General disorders) | 1 (1)
Intermittent headaches (Nervous system disorders) | 1 (1)
Intestinal virus (Infections and infestations) | 1 (1)
Irritation on sensor site (General disorders) | 1 (1)
Iv site pain (General disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Left leg cellulitis (Infections and infestations) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Mononucleosis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pain (General disorders) | 1 (1)
Periodontal infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Severe hyperglycemia (Metabolism and nutrition disorders) | 13 (17)
Sinus infection (Infections and infestations) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach flu (Infections and infestations) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Type 4 skin hypersensitivity (Immune system disorders) | 1 (1)
Upper respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Uti (Infections and infestations) | 2 (2)
Viral illness (Infections and infestations) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days